CLINICAL TRIAL: NCT05803798
Title: Combined Treatment With Pulsed Light and Photobiomodulation Before Laser Refractive Surgery
Acronym: TEBELID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC22.0190
Record Dates: First submitted 2023-03-21; First posted 2023-04-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye; Dry Eye After LASIK-Laser in Situ Keratomileusis
Keywords: dry eye; laser refractive surgery; smile; lasik; presbylasik; photorefractive keratectomy; intense-pulsed light; low-level-light therapy; photobiomodulation
MeSH Terms: conditions — Dry Eye Syndromes; Smiling

STUDY DESIGN:
Intervention Model Description: Treatment group = LLLT+IPL (EYE-LIGHT) before laser refractive surgery
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Active Comparator): preventive treatment by IPL+LLLT with EYE-LIGHT, Espansione group
  Interventions: Device: IPL+LLLT
- standard (No Intervention): non preventive treatment by IPL+LLLT with EYE-LIGHT, Espansione group = standard care

INTERVENTIONS:
Device: IPL+LLLT — preventive treatment by IPL+LLLT (EYE-LIGHT) before laser refractive surgery
  Arms: treatment

SUMMARY:
Laser corneal refractive surgery is a widely adopted approach for correcting refractive errors, but postoperative dry eye remains a common side effect. Intense Pulsed Light (IPL) and Low-Level Light Therapy (LLLT) are two emerging treatments that have shown potential in managing dry eye disease. However, their role as a prophylactic treatment in patients without pre-existing symptomatic dry eye undergoing refractive surgery has not been explored.

DETAILED DESCRIPTION:
monocentric, randomized, simple bling, controlled study

ELIGIBILITY:
Patients eligible for laser corneal refractive surgery (FS-LASIK, SMILE®, or PRK) who meet the inclusion criteria will be enrolled.

Exclusion criteria include age < 18 and contraindications to IPL or LLLT (e.g., pregnancy, lactation, migraine, epilepsy, palpebral or periocular lesion, photosensitive drugs, cardiac pacing system or implantable cardiovertor defibrillator, Fitzpatrick phototypes V and VI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
French version of Ocular Surface Disease Index (OSDI) score | 1 month post-operative
  The OSDI questionnaire measures frequency of symptoms, environmental triggers and vision related quality of life.
  OSDI values range from 0 to 100. A score between 13 and 22 excluded indicates a medium intensity eye dryness. A score between 22 and 33 indicated a moderate intensity eye dryness. A score above 33 indicates a severe eye dryness.

SECONDARY OUTCOMES:
Evolution of Fluorescein Break-up Time (FBUT) over the 6 first months post-operative | 6 months post-operative
  Sodium fluorescein eye drops is instilled in the eye to enhance visibility of the tear film measure tear film breakup time is. Selected cut-off value is 10 seconds. A score below 10 seconds favors dry eye.
Evolution of Schirmer I test over the 6 first months post-operative | 6 months post-operative
  The Schirmer I test, used without anesthesia, provides an estimation of stimulated reflex. Cut-off value used is <= 10 mm / 5 minutes.
Evolution of Meibomian Gland Dropout over the 6 first months post-operative | 6 months post-operative
  Meibomian Gland Dropout: Evaluated via infrared images using LipiView™ II (Quantel Medical) and graded using the Gestalt Grading Scale (GGS), which scores meibomian gland loss on a scale from 1 (no loss) to 4 (>75% loss).
Evolution of the Oxford score over the 6 first months post-operative | 6 months post-operative
  The Oxford score is composed of 0 to V grades, dependent on intensity of punctate staining displayed.
  pictorially across a combination of the cornea and conjunctiva.
Evolution of visual acuity over the 6 first months post-operative | 6 months post-operative
  Visual acuity measured preoperatively (corrected) and postoperatively (uncorrected) using the Early Treatment of Diabetic Retinopathy Study (ETDRS) scale at 4 meters. Visual acuity is scored by adding 30 to the total number of letters read correctly at 4 meters
Evolution of the French version of Ocular Surface Disease Index (OSDI) score over the 6 first months post-operative | 6 months post-operative
  The OSDI questionnaire measures frequency of symptoms, environmental triggers and vision related quality of life.
  OSDI values range from 0 to 100. A score between 13 and 22 excluded indicates a medium intensity eye dryness. A score between 22 and 33 indicated a moderate intensity eye dryness. A score above 33 indicates a severe eye dryness.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice COCHENER-LAMARD, MD, PhD, Principal Investigator — Universitary Hospital of Brest
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified (coded/pseudonymised) individual participant data from the TEBeLiD randomized trial that underlie the primary and secondary publications/final study report. Dataset includes baseline demographics/clinical characteristics, randomization group, procedural variables, follow-up outcomes (e.g., F-OSDI/OSDI, tear film break-up time, corneal staining/Oxford score, Schirmer test, meibomian gland assessment/meibography), adverse events, and protocol deviations. A data dictionary and variable coding will be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital (CHU de Brest). Requests must include a research proposal and analysis plan (and ethics approval/exemption if applicable). Approved requestors will be required to sign and comply with a data access/data use agreement (no re-identification; secure storage; no onward sharing; acknowledgement/citation of TEBeLiD investigators). Data will be provided via secure transfer or controlled-access environment.

REFERENCES:
- [Background] Dartt DA. Neural regulation of lacrimal gland secretory processes: relevance in dry eye diseases. Prog Retin Eye Res. 2009 May;28(3):155-77. doi: 10.1016/j.preteyeres.2009.04.003. Epub 2009 Apr 17. PMID 19376264
- [Background] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Background] Tashbayev B, Yazdani M, Arita R, Fineide F, Utheim TP. Intense pulsed light treatment in meibomian gland dysfunction: A concise review. Ocul Surf. 2020 Oct;18(4):583-594. doi: 10.1016/j.jtos.2020.06.002. Epub 2020 Jul 3. PMID 32629039
- [Background] Cote S, Zhang AC, Ahmadzai V, Maleken A, Li C, Oppedisano J, Nair K, Busija L, Downie LE. Intense pulsed light (IPL) therapy for the treatment of meibomian gland dysfunction. Cochrane Database Syst Rev. 2020 Mar 18;3(3):CD013559. doi: 10.1002/14651858.CD013559. PMID 32182637
- [Background] McDonald M, Patel DA, Keith MS, Snedecor SJ. Economic and Humanistic Burden of Dry Eye Disease in Europe, North America, and Asia: A Systematic Literature Review. Ocul Surf. 2016 Apr;14(2):144-67. doi: 10.1016/j.jtos.2015.11.002. Epub 2015 Dec 28. PMID 26733111
- [Background] Stapleton F, Alves M, Bunya VY, Jalbert I, Lekhanont K, Malet F, Na KS, Schaumberg D, Uchino M, Vehof J, Viso E, Vitale S, Jones L. TFOS DEWS II Epidemiology Report. Ocul Surf. 2017 Jul;15(3):334-365. doi: 10.1016/j.jtos.2017.05.003. Epub 2017 Jul 20. PMID 28736337
- [Background] Gomes JAP, Azar DT, Baudouin C, Efron N, Hirayama M, Horwath-Winter J, Kim T, Mehta JS, Messmer EM, Pepose JS, Sangwan VS, Weiner AL, Wilson SE, Wolffsohn JS. TFOS DEWS II iatrogenic report. Ocul Surf. 2017 Jul;15(3):511-538. doi: 10.1016/j.jtos.2017.05.004. Epub 2017 Jul 20. PMID 28736341
- [Background] Denoyer A, Landman E, Trinh L, Faure JF, Auclin F, Baudouin C. Dry eye disease after refractive surgery: comparative outcomes of small incision lenticule extraction versus LASIK. Ophthalmology. 2015 Apr;122(4):669-76. doi: 10.1016/j.ophtha.2014.10.004. Epub 2014 Nov 22. PMID 25458707
- [Background] Kim TI, Alio Del Barrio JL, Wilkins M, Cochener B, Ang M. Refractive surgery. Lancet. 2019 May 18;393(10185):2085-2098. doi: 10.1016/S0140-6736(18)33209-4. PMID 31106754